CLINICAL TRIAL: NCT03224000
Title: Bayesian Phase II Trial of Magnetic Resonance Imaging Guided Radiotherapy Dose Adaptation in Human Papilloma Virus Positive Oropharyngeal Cancer
Brief Title: Trial of Magnetic Resonance Imaging Guided Radiotherapy Dose Adaptation in Human Papilloma Virus Positive Oropharyngeal Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2015-0851; NCI-2018-01109 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2017-07-14; First posted 2017-07-21 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Malignant Neoplasms of Lip Oral Cavity and Pharynx; Oropharyngeal Cancer
Keywords: Malignant neoplasms of lip oral cavity and pharynx; Oropharyngeal Cancer; Human papilloma virus positive; HPV+; Squamous cell carcinoma of the oropharynx; Squamous cell carcinoma of the tonsil; Squamous cell carcinoma of the base of tongue; Squamous cell carcinoma of the soft palate; Squamous cell carcinoma of the oropharyngeal walls; Magnetic Resonance Imaging Guided Radiotherapy; Standard of Care Radiotherapy Planning; Radiation Therapy; Intensity modulated radiotherapy; IMRT; Modified Barium Swallow; MBS; Swallowing questionnaire; The M.D. Anderson Dysphagia Inventory (MDADI); Symptom questionnaire; The M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN); Video-Strobe Procedure
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck; Head and Neck Neoplasms | interventions — Radiotherapy, Intensity-Modulated; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- MRI Guided Intensity Modulated Radiotherapy (IMRT) (Experimental): Modified barium swallow (MBS) performed at baseline and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Swallowing questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Symptom questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Video-strobe procedure performed at baseline, at week 3 during radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  IMRT planned with MRI guidance. Participants receive an individualized prescription of up to 70 Gy in 33 fractions with radiation therapy (RT) given once daily, 5 days a week, over 6 weeks and 3 days.
  Interventions: Procedure: Modified Barium Swallow (MBS); Behavioral: Swallowing Questionnaire; Behavioral: Symptom Questionnaire; Procedure: Video-Strobe Procedure; Procedure: MRI Guided Intensity Modulated Radiotherapy (IMRT) Planning; Radiation: Intensity Modulated Radiotherapy (IMRT)
- Standard-of-Care Intensity Modulated Radiotherapy (IMRT) (Active Comparator): Modified barium swallow (MBS) performed at baseline and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Swallowing questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Symptom questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Video-strobe procedure performed at baseline, at week 3 during radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  IMRT planned by standard-of-care. Participants receive an individualized prescription of up to 70 Gy in 33 fractions with radiation therapy (RT) given once daily, 5 days a week, over 6 weeks and 3 days.
  Interventions: Procedure: Modified Barium Swallow (MBS); Behavioral: Swallowing Questionnaire; Behavioral: Symptom Questionnaire; Procedure: Video-Strobe Procedure; Procedure: Standard-of-Care Intensity Modulated Radiotherapy (IMRT) Planning; Radiation: Intensity Modulated Radiotherapy (IMRT)

INTERVENTIONS:
Procedure: Modified Barium Swallow (MBS) — Modified barium swallow (MBS) performed at baseline and at 6 months, 2 years, and 5 years after finishing radiation therapy.
Behavioral: Swallowing Questionnaire — Swallowing questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Other Names: The M.D. Anderson Dysphagia Inventory (MDADI)
Behavioral: Symptom Questionnaire — Symptom questionnaire completed at baseline, every week while receiving radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
  Other Names: The M.D. Anderson Symptom Inventory for Head and Neck Cancer (MDASI-HN)
Procedure: Video-Strobe Procedure — Video-strobe procedure to check vocal cords performed at baseline, at week 3 during radiation therapy, and at 6 months, 2 years, and 5 years after finishing radiation therapy.
Procedure: MRI Guided Intensity Modulated Radiotherapy (IMRT) Planning — IMRT planned with MRI guidance.
  Arms: MRI Guided Intensity Modulated Radiotherapy (IMRT)
Procedure: Standard-of-Care Intensity Modulated Radiotherapy (IMRT) Planning — IMRT planned by standard-of-care.
  Arms: Standard-of-Care Intensity Modulated Radiotherapy (IMRT)
Radiation: Intensity Modulated Radiotherapy (IMRT) — Participants receive an individualized prescription of up to 70 Gy in 33 fractions with radiation therapy (RT) given once daily, 5 days a week, over 6 weeks and 3 days.
  Other Names: Radiation therapy; XRT

SUMMARY:
The goal of this clinical research study is to compare the use of MRI simulations to plan different doses of intensity modulated radiotherapy (IMRT) to the standard IMRT dose in patients with low risk human papilloma virus positive oropharyngeal cancer.

This is an investigational study. MRI simulations and radiation therapy are delivered using FDA-approved and commercially available methods. The use of MRI imaging to plan the dose is investigational.

Up to 90 participants will be enrolled in this study. All will take part at MD Anderson.

DETAILED DESCRIPTION:
Baseline Visit:

If you are found to be eligible to take part in this study and agree, you will have a baseline visit. The following tests and procedures will be performed:

* You will have a hearing test.
* You will have a dental exam. During this exam, your saliva flow will be measured and you will be checked for lockjaw.
* Your swallowing function will be tested with a special type of x-ray called a modified barium swallow (MBS). During the test, you will eat and drink foods and liquids mixed with a "contrast" chemical called barium that will make your throat more visible in the x-rays. A special x-ray tube will be connected to a television screen to allow the doctor to watch the foods and liquids pass from your mouth and down your throat.
* You will complete a questionnaire about swallowing that should take about 5 minutes to complete.
* You will have a video-strobe procedure to check your vocal cords. To perform a video-strobe procedure, a small camera will be inserted into the throat through your nose or mouth. You will be awake for this procedure and the study staff will give you the option of receiving a numbing spray for your nose and/or throat.
* Photos of the inside of your mouth will be taken to check for mouth sores.
* You will fill out questionnaires about your quality of life, work status, medical history, smoking status, and any symptoms you may have. Completing these questionnaires should take about 10-15 minutes.

Study Groups:

If you are among the first 15 patients enrolled in the study, you will be in Group 1.

If you join the study after the first 15 patients have enrolled, you will be randomly assigned (as a flip of a coin) to 1 of 2 study groups. This is done because no one knows if one study group is better, the same, or worse than the other group.

* If you are in Group 1, an MRI will be used to plan your IMRT.
* If you are in Group 2, you will receive standard-of-care IMRT.

Length of Study Participation:

No matter which group you are in, you may continue receiving radiation therapy for up to 6 ½ weeks. You will no longer be able to take part in this study if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your overall participation on the study will be over after 5 years.

Treatment Planning and Schedule:

You will receive a standard CT simulation which will cover your head and neck for treatment planning. You will also have a PET-CT to check the status of the disease and for treatment planning purposes.

If you are among the first 15 participants or are in Group 1, you also will have an MRI simulation for treatment planning purposes.

All groups will then receive radiation therapy 1 time each day, 5 days a week (Monday through Friday) for up to 33 treatments (about 6 ½ weeks).

Study Visits:

Every week while you are receiving radiation therapy:

* You will have a physical exam.
* Blood (about 1-2 tablespoons) will be drawn for routine tests.
* You will fill out the same questionnaires as before.
* You will have an MRI.

At Weeks 3 and 6:

* Photos of the inside of your mouth will be taken to check for mouth sores.
* You will have a dental exam.

If you are among the first 15 participants or are in Group 1, you will also have the MRI simulation at the end of Weeks 1, 2, 3, and 4 of treatment.

Six (6) weeks after finishing radiation therapy, you will complete the same questionnaires as before.

Within 8-12 weeks after finishing radiation therapy:

* Photos of the inside of your mouth will be taken to check for mouth sores.
* You will have a hearing test.
* If you are among the first 15 participants or are in Group 1, you will have an MRI simulation.

Six (6) months, 1 year, and 2 years after finishing radiation therapy:

* You will fill out the same questionnaires as before.
* You will have a mouth exam to check your swallowing function.
* Photos of the inside of your mouth will be taken to check for mouth sores.
* You will fill out the same questionnaires as before.
* You will have a video-strobe procedure to check your vocal cords.
* At 1 year only, you will have a dental exam and an MBS exam to test your swallowing function.
* At 1 year and 2 years only, you will also have a hearing test.

Three to six (3-6) months, 1 year, and 18-24 months after finishing radiation therapy:

* You will have an MBS exam to test your swallowing function.
* You will fill out the same questionnaires as before.
* You will have the video-strobe procedure to check your vocal cords.

Two (2) years after finishing radiation therapy and if the disease gets worse, blood (about 3 teaspoons) will be drawn for circulating tumor cells (CTCs). This is a test of how many tumor cells are in the blood.

Five (5) years after finishing radiation therapy, you will have an MBS exam to test your swallowing function and will complete the same questionnaires as before.

If the doctor thinks it is needed during follow-up, you will have a tumor biopsy for tumor marker testing and a CT scan, MRI scan and/or PET/CT scan to check the status of the disease.

Follow-Up Calls:

During the 8-12 weeks while you are recovering from treatment, you will be called or emailed by an automated system every 2 weeks.

This will be to remind you to fill out a web-based form that asks about any side effects you may have had. Completing the form should take about 10-15 minutes each time.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy proven diagnosis of squamous cell carcinoma of the oropharynx (tonsil, base of tongue, soft palate, or oropharyngeal walls). Clinical evidence should be documented, and may consist of imaging, endoscopic evaluation, palpation, and should be sufficient to estimate the size of the primary for purposes of T staging.
* Age ≥18 years
* Clinical stage T1-3, N0-2 (AJCC, 8th ed.), with no distant metastases, based on routine staging workup.
* Positive for HPV by p16 IHC or ISH
* Lifetime pack-year history of <10 years, currently non-smoking for at least 5 years.
* No head and neck surgery of the primary tumor or lymph nodes except for incisional or excisional biopsies.
* No retropharyngeal nor level IV (or lower) lymphadenopathy (i.e. nodes in level I-III only)
* Eastern Cooperative Oncology Group (ECOG) = 0, 1, or 2.
* Dispositioned to photon/proton radiotherapy +/- chemotherapy
* For females of child-bearing age, a negative pregnancy test

Exclusion Criteria:

* Patients who have undergone definitive resection of their primary or nodal disease as well as any chemotherapy or radiation therapy for their HNSCC.
* Pregnant or breast-feeding females
* Clinically significant uncontrolled major cardiac, respiratory, renal, hepatic, gastrointestinal or hematologic disease but not limited to:
* Symptomatic congestive heart failure, unstable angina, or cardiac dysrhythmia not controlled by pacer device
* Myocardial infarction within 3 months of registration
* Contraindications to MR imaging (e.g. implanted metallic prostheses, defibrillators, stimulators, pacemakers, or neurotransmitters) per institutional policy on management of patients with internal and external medical devices.
* History of claustrophobia
* Having an estimated glomerular filtration rate (GFR) < 40ml/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2018-01-17 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Locoregional Control | 6 months post radiation therapy
  Relapse defined as reappearance of tumor after complete response. If possible, relapse confirmed by biopsy.
Composite Dysphagia Outcome Determined by PEG Tube Dependence at Last Follow-Up | 6 months post radiation therapy
  Composite dysphagia outcome calculated based on objective measurements of severe dysphagia.
  These include: 1) PEG tube dependence at last follow-up; 2) trace or frank aspiration seen on modified barium swallow study; 3) diagnosis of aspiration pneumonia; 4) presence of pharyngoesophageal structure on modified barium swallow study or endoscopy with subsequent need for dilation.
Composite Dysphagia Outcome Determined by Trace or Frank Aspiration Seen on Modified Barium Swallow Study | 6 months post radiation therapy
  Composite dysphagia outcome calculated based on objective measurements of severe dysphagia.
Composite Dysphagia Outcome Determined by Diagnosis of Aspiration Pneumonia | 6 months post radiation therapy
  Composite dysphagia outcome calculated based on objective measurements of severe dysphagia.
Composite Dysphagia Outcome Determined by Presence of Pharyngoesophageal Structure on Modified Barium Swallow Study | 6 months post radiation therapy
  Composite dysphagia outcome calculated based on objective measurements of severe dysphagia.
Composite Dysphagia Outcome Determined by Presence of Pharyngoesophageal Structure on Endoscopy with Subsequent Need for Dilation | 6 months post radiation therapy
  Composite dysphagia outcome calculated based on objective measurements of severe dysphagia.

SECONDARY OUTCOMES:
Overall Survival | Start of treatment up to 5 years
  Overall survival, calculated as time from diagnosis to either death or last follow-up, with death serving as an event and all others censored.
Progression-Free Survival | Start of treatment up to 5 years
  Progression-free survival, calculated as time from diagnosis to either death or detection of recurrent disease after an interval without radiographic of clinically evident disease (whichever is earlier), with death or recurrence detection serving as an event and all others censored.
Distant Metastasis-Free Survival | Start of treatment up to 5 years
  Distant metastasis-free survival, calculated as time from diagnosis to either death or detection of disease outside of the head and neck after an interval without radiographic of clinically evident disease (whichever is earlier), with death or metastasis detection serving as an event and all others censored.
Patient Reported Outcome (PRO) Measures of Symptoms Using MD Anderson Symptom Inventory (MDASI) | Baseline up to 2 years after radiation therapy
  Patient Reported Outcome (PRO) measures of symptoms using MD Anderson Symptom Inventory (MDASI)
Physician-Reported Toxicity | Weekly during radiation therapy up to 2 years after radiation therapy
  Physician-reported toxicity, defined as any grade 3-4 adverse events using Common Terminology Criteria for Adverse Events (CTCAE)-4.0.
Patient Reported Outcome (PRO) Measures of Symptoms Using MD Anderson Dysphagia Inventory (MDADI) | Baseline up to 2 years after radiation therapy
Patient Reported Outcome (PRO) Measures of Symptoms Using FACT-HN | Baseline up to 2 years after radiation therapy
Patient Reported Outcome (PRO) Measures of Symptoms Using Xerostomia and Health Questionnaire (EQ-5D-3L) | Baseline up to 2 years after radiation therapy
Patient Reported Outcome (PRO) Measures of symptoms Using Performance Status Scale-HN | Baseline up to 2 years after radiation therapy
Patient Reported Outcome (PRO) Measures of symptoms Using Work Productivity and Activity Impairment Questionnaire | Baseline up to 2 years after radiation therapy

CONTACTS AND LOCATIONS:
Overall Officials: Clifton Fuller, MD, PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Bahig H, Yuan Y, Mohamed ASR, Brock KK, Ng SP, Wang J, Ding Y, Hutcheson K, McCulloch M, Balter PA, Lai SY, Al-Mamgani A, Sonke JJ, van der Heide UA, Nutting C, Li XA, Robbins J, Awan M, Karam I, Newbold K, Harrington K, Oelfke U, Bhide S, Philippens MEP, Terhaard CHJ, McPartlin AJ, Blanchard P, Garden AS, Rosenthal DI, Gunn GB, Phan J, Cazoulat G, Aristophanous M, McSpadden KK, Garcia JA, van den Berg CAT, Raaijmakers CPJ, Kerkmeijer L, Doornaert P, Blinde S, Frank SJ, Fuller CD. Magnetic Resonance-based Response Assessment and Dose Adaptation in Human Papilloma Virus Positive Tumors of the Oropharynx treated with Radiotherapy (MR-ADAPTOR): An R-IDEAL stage 2a-2b/Bayesian phase II trial. Clin Transl Radiat Oncol. 2018 Aug 24;13:19-23. doi: 10.1016/j.ctro.2018.08.003. eCollection 2018 Nov. PMID 30386824
- See also: M D Anderson Cancer Center — http://www.mdanderson.org